CLINICAL TRIAL: NCT03057132
Title: A Pilot Study Evaluating the Use of 3M Cavilon Advanced Skin Protectant in the Management of Damaged Skin Around an Ostomy, Drain or Fistula
Brief Title: Use of 3M Cavilon Advanced Skin Protectant in the Management of Damaged Skin Around an Ostomy, Drain or Fistula
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment of patients
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CLIN-PROT-ICH-US-05-274494
Record Dates: First submitted 2017-01-09; First posted 2017-02-17 (Actual); Results first posted 2019-06-04 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Ostomy

STUDY DESIGN:
Masking Description: Open label no masking required
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cavilon Advanced Skin Protectant (Experimental): Cavilon Advanced Skin Protectant
  Interventions: Device: Cavilon Advanced Skin Protectant

INTERVENTIONS:
Device: Cavilon Advanced Skin Protectant — Cavilon Advanced Skin Protectant

SUMMARY:
The objective of this pilot study is to evaluate the feasibility, safety and efficacy of 3M™ Cavilon™ Advanced Skin Protectant when used in the management of damaged skin exposed to caustic body fluids from an ostomy, drain site or fistula.

DETAILED DESCRIPTION:
This is a pilot study evaluating the product, 3M™ Cavilon™ Advanced Skin Protectant, for the management of skin around an ostomy, drain and/or fistula. All subjects will receive the product for up to 14 days. The primary site must have red skin with breakdown (i.e. skin erosion and denudation or denudation of skin alone). Secondary sites can have red skin with or without breakdown. Product will be applied twice/week or more frequently if additional applications are needed due to leakage, skin irritation or standard of care. Skin assessments (including photography) will be completed at baseline and at all follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Is the subject 18 years of age or older?
2. Does the subject have red skin with breakdown (i.e. skin erosion and denudation or denudation of skin alone) at the primary site of an ostomy, drain and/or fistula?
3. Is the subject willing to have photographs taken of their skin and permit use of photographs in potential publication?
4. Is the subject willing to release rights to 3M for the use of the photos?
5. Is there a reasonable expectation that the subject will be in the hospital or available for follow-up visits during the 14 day study period?
6. Has the subject signed an Institutional Review Board-approved informed consent/assent document and authorized the use and disclosure of protected health information?

Exclusion Criteria:

1. If female, is the subject pregnant or breast feeding or has she given birth within the 3 weeks preceding the screening visit?
2. Does the subject have a known allergy to acrylates or cyanoacrylates?
3. Does the subject have a preexisting skin disease on the areas affected that may make skin assessments for this study difficult?
4. Does the skin area affected require treatment with a concomitant medication or product?
5. Has the subject received antifungal powders in the area affected within 24 hours prior to enrollment?
6. Has the subject received cyanoacrylate based skin protectant (such as Marathon) within 72 hours prior to enrollment?
7. Does the subject have any medical condition that in the opinion of the investigator should exclude him/her from participating in the study?
8. Has the subject been enrolled in any investigational study where product was applied to proposed study sites within 30 days of the screening visit?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cooper, MD, Study Director — 3M
Locations (1):
- Eastern Regional Medical Center, Inc., Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cavilon Advanced Skin Protectant: Single topical application of Cavilon Advanced Skin Protectant to skin around the ostomy
Period: Overall Study
Arm/Group | Cavilon Advanced Skin Protectant
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One male subject completed this study. The subject was a 63 year old white male.
Groups:
- Cavilon Advanced Skin Protectant: Cavion Advanced Skin Protectant was applied to one male subject.
Arm/Group | Cavilon Advanced Skin Protectant
Number analyzed (Participants) | 1
Age, Customized [Number; unit: years]
  Age of Subject | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Number of participants [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent of Epidermal Skin Loss at the Primary Site Assessed
Description: The primary endpoint is the improvement of denuded skin (defined as clinical improvement from the baseline skin assessment) of the primary site of interest (ostomy).
  The primary response was the percent of skin at primary site of interest with epidermal loss observed at baseline and at 3 days post product application.
Time Frame: Baseline, 3 days
Population: One application of Cavilon Advanced Skin Protectant was applied around the ostomy site. Skin was assessed at baseline and at 3 days after product application.
Measure: Number; unit: Percentage of epidermal skin loss
Groups:
- Cavilon Advanced Skin Protectant: Assessed area around an ostomy and estimated the percentage of skin that was normal, intact with pink/redness, and had epidermal loss (denuded).
Arm/Group | Cavilon Advanced Skin Protectant
Number analyzed (Participants) | 1
Percentage of epidermal skin loss
  Baseline % epidermal loss | 10
  Day 3 % epidermal loss | 0

2. Primary Outcome: Pain Scores at the Primary Site Assessed
Description: Improvement in pain from baseline to the end of the study. The Wong-Baker FACES® Pain Visual Analog Pain Scale was used to assess pain at each time point. Pain was assessed on a 0 (no pain) to 10 (worst pain) grading scale. Lower score is better.
Time Frame: Baseline, 3 days
Population: Pain was rated during and after cleansing at baseline and at Day 3, and during and after product application at baseline.
Measure: Number; unit: units on a scale
Groups:
- Cavilon Advanced Skin Protectant: Pain was rated during and after cleansing at baseline and at Day 3. Pain was rated during and after product application.
Arm/Group | Cavilon Advanced Skin Protectant
Number analyzed (Participants) | 1
units on a scale
  Baseline Pain During Cleaning | 2
  Baseline Pain After Cleaning | 2
  Baseline Pain During Application | 2
  Baseline Pain After Application | 0
  Day 3 Pain During Cleaning | 0
  Day 3 Pain After Cleaning | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected through study completion (3 days).
Description: There were no adverse events during the study.
Groups:
- Cavilon Advanced Skin Protectant: Cavilon Advanced Skin Protectant-single arm study
Arm/Group | Cavilon Advanced Skin Protectant
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early termination due to enrollment issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT03057132/Prot_SAP_000.pdf